CLINICAL TRIAL: NCT01892891
Title: A Double-Blind, Randomized, Placebo-Controlled, Sequential, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral Doses of VBY-036 in Healthy Subjects
Brief Title: Safety Study of VBY-036 in Healthy Volunteers After 7 Days of Oral Dosing
Acronym: VBY036P1B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virobay Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: VBY-036-002
Record Dates: First submitted 2013-07-01; First posted 2013-07-08 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: Healthy; Subjects; Safety; Tolerability; VBY036; maximum; pharmacodynamic; pharmacokinetic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VBY-036 (Experimental): VBY-036 30 mg, 100 mg, 300 mg, 600 mg, or 900 mg
  Interventions: Drug: VBY-036
- Placebo comparator (Placebo Comparator): Placebo

INTERVENTIONS:
Drug: VBY-036 — Cathepsin S inhibitor
  Arms: VBY-036

SUMMARY:
VBY-036 may treat or prevent nerve pain. This study aims to find the highest safe and tolerable dose of VBY-036 in healthy volunteers. Volunteers will be randomly selected to receive either a placebo or VBY-036 (30, 100, 300, 600 or 900 mg) once daily for seven days in a row.

DETAILED DESCRIPTION:
Detailed description is noted in Brief Summary.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-60 years old
* Screening body mass index between 18-32 kg/m2
* Good health, no clinically significant findings in medical history, 12-lead ECG, & vital signs;
* Clinical lab evaluations (Chem panel [fasted at least 8 hrs], CBC, HbA1c & UA in reference range for test lab (unless deemed not clinically significant);
* Negative test for drugs of abuse at Screening & at Check-in (includes alcohol);
* Negative hepatitis, HIV & TB screens;
* Females non-pregnant, non-lactating, & either postmenopausal for at least 1 year, surgically sterile for at least 90 days prior to Check-in, or agree to use from the time of consent until 90 days after Study Completion an effective form of contraception. For all females, a pregnancy test result must be negative at Screening & Check-in.
* Males will be sterile or agree to use from Check-in until 90 days following discharge an effective method of contraception.
* Able to comprehend & willing to sign Informed Consent Form

Exclusion Criteria:

* Females pregnant or nursing, or childbearing potential but unwilling to use contraception.
* History of renal or hepatic impairment; stomach or intestinal surgery or resection, malabsorption syndrome, cholecystectomy, or gastro-intestinal dysfunction that would alter absorption &/or excretion of orally administered drugs (appendectomy or hernia repair allowed);
* Anemia (hemoglobin <11.5 g/dL for females; < 13 g/dL for males) or blood donation within 8 weeks of Check-in;
* Plasma donation within 4 weeks of Check-in;
* History of alcoholism or drug addiction within 6 months to Check-in;
* Use of drugs of abuse or prescription drugs for recreational use 6 months prior to Check-in;
* Use of any tobacco-containing or nicotine-containing products 6 months prior to Check-in & during study;
* Participation in another drug trial 30 days of Check-in (within 8 weeks if previous investigational drug has immunomodulary effects, other than cathepsin S inhibition);
* History or clinical manifestations of metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, urological, neurological, or psychiatric disorders
* History of hypersensitivity or allergies to any drug compound
* History or presence of abnormal ECG
* Laboratory abnormality deemed clinically significant;
* Use of or inability to discontinue any prescription medications/products 14 days prior to Check-in & during study;
* Use of certain over-the-counter, non-prescription preparations are permitted up to 3 days before first dose;
* Use of alcohol-containing, grapefruit-containing, star fruit containing foods or beverages or "energy drinks" 72 hours to Check-in & during study;
* Poor peripheral venous access;
* Receipt of blood products 6 months to Check-in
* Subjects with history of Gilbert's Syndrome;
* Strenuous activities 48 hours to Check-in
* Illness 5 days to drug administration
* Any acute or chronic condition

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Highest safe and tolerated VBY-036 dose | 7 days of dosing
  Single dose of VBY-036 given daily for 7-days in a row for each cohort in an ascending manner.
  Cohort B1 with 30 mg dose or placebo; Cohort B2 with 100 mg dose or placebo; Cohort B3 with 300 mg dose or placebo; Cohort B4 with 600 mg dose or placebo; Cohort B5 with 900 mg dose or placebo

SECONDARY OUTCOMES:
Confirmation of cathepsin-S inhibition | 7 days
  Based on the accumulation of Iip 10 and/or cathepsin S protein levels

OTHER OUTCOMES:
The blood level of VBY-036 | 7 days
  The blood level of VBY-036 across the dose range of 30 mg to 900 mg

CONTACTS AND LOCATIONS:
Overall Officials: David B. Karpf, MD, Study Director — Virobay Inc.
Locations (1):
- Covance Evansville, Evansville, Indiana, United States